CLINICAL TRIAL: NCT04646161
Title: Prostaglandins Use Before Mirena IUD Insertion in Prev CS Women During Lactational Amenorrhea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany saad, assisstant professor, Cairo University
Other Study IDs: professor
Record Dates: First submitted 2020-11-07; First posted 2020-11-27 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: to Study the Estimate Difficulty of Insertion Mirena IUD With Use of Prostaglandins
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- prostaglandins before iud insertion group: this group will receive 200 mcg prostaglandins in form of misoprostol 2 hrs before mirena iud insertion
  Interventions: Drug: Misoprostol
- placebo group: this group will receive placebo tablet before mirena iud insertion

INTERVENTIONS:
Drug: Misoprostol — misoprostol 200 mcg will be given sublingual 2 hrs before mirena iud insertion
  Groups: prostaglandins before iud insertion group

SUMMARY:
This is a prospective randomized controlled study to determine the effect of prostaglandin intake before Mirena IUD insertion It was conducted at the Department of Obstetrics & Gynecology, Kasr El-Ainy Teaching Hospital, Faculty of Medicine, Cairo University,

DETAILED DESCRIPTION:
The study aiming to measure the estimate difficulty of insertion of the Mirena IUD by using prostaglandins 2 hours before the procedure and the effect of prostaglandins to make this procedure easy with other side effects and complications as bleeding perforation, nausea, vomiting, failure of insertion and comparing them with a placebo group who didn't receive prostaglandins

ELIGIBILITY:
Inclusion Criteria:

* 1- Women in lactational amenoeehea with pregnancy test negative 2- Women who had caesarean section within 6 monthes of IUD insertion 3- No medical disorders

Exclusion Criteria:

* 1- Women in regular menses 2- Medical disorders 3- Nulligravida or muligravida with NVD 4- Women with history of Previous CS more than one CS 5- Any congenital uterine anomalies, fibroids and adenomysis 6- Chronic pelvic pain 7- Intrauterine adhesions 8- Spasmodic dysmenohrrea 9- Allergy to misoprostol

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: female patients during the lactational amenorrhea who undergo Mirena IUD insertion after had been delivered by CS within 6 monthes
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Difficulty of insertion of Mirena IUD by using the Ease of Insertion score graduated as VAS like scale | During the intervention
  By using the visual analogue score

SECONDARY OUTCOMES:
cervical dilataion < 4 mm | During the intervention
  need for cervical dilatation to pass the IUD
Pain at insertion according to VAS | During the intervention
  By using the visual analogue score
Subjective sensation of satisfaction graduated as VAS like scale | During the intervention
  By using the visual analogue score like system
side effects during IUD insertion: bleeding, vasovagal reaction, cramps, nausea, perforation, vomiting | During the intervention
  Bleeding by using the soaked bads
side effects after 24 hrs of IUD insertion: nausea, vomiting, cramps and hyperthermia | During the first 24 hours
side effects after 30 days of IUD insertion: spotting, cramps, acute PID and expulsion | After 30 days of intervention
Duration of insertion(min) | During the intervention
  From start of procedure till removing the speculum

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided